CLINICAL TRIAL: NCT05915559
Title: Outpatient Management of Tonsillectomy in Adults
Acronym: AMYAMBU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0115
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Tonsillectomy; Pain; Ambulatory
Keywords: Tonsillectomy; Pain; ambulatory
MeSH Terms: conditions — Pain | interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tonsillectomy (Experimental)
  Interventions: Procedure: Tonsillectomy; Other: daily follow-up

INTERVENTIONS:
Procedure: Tonsillectomy — Tonsillectomy
Other: daily follow-up — daily follow-up of clinical parameters (pain, feeding) and analgesia adapted to the pain

SUMMARY:
Tonsillectomy is a frequent surgical procedure in the ENT specialty but it can be a source of postoperative pain that can be important. These pains complicate the intake of food and in particular the intake of analgesic drugs per os and require the prolongation of the hospitalization in order to continue an intravenous analgesia. The aim is to set up a protocol for ambulatory care of adult tonsillectomies. Then, it would allow an improvement of the postoperative quality of life for the patient, who prefers a quicker return home.The study aims to allow patients to come back home early after tonsillectomies with intravenous analgesia. Pain, feeding and quality of life will be evaluated regularly through an application called MAELA during a few days after surgery. They will also be evaluated by nurses coming via providers.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a tonsillectomy defined in the French recommendations
* Age between 18 and 60 yo
* Providing free and informed consent to participate
* Having a smartphone able to process MAELA application
* Affiliation to french social security

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients EVA score less or equal at 3 | day 1
  EVA score is a pain scale from 0 to 10. 10 is the highest pain level.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No